CLINICAL TRIAL: NCT05588518
Title: Randomized Clinical Trial and Comparison of Propolis With Sodium Fluoride and Acidulated Phosphate Fluoride Using Iontophoresis as a Treatment for Cervical Dentin Hypersensitivity
Brief Title: Propolis as a Treatment for Cervical Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Raghavendra Reddy Nagate, Assistant Professor, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB/KKUCOD/ETH/2018-19/112
Record Dates: First submitted 2022-10-15; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Dental Root Sensitivity
Keywords: Dental calculus; Dentine sensitivity; Gingival recession
MeSH Terms: conditions — Dental Calculus; Dentin Sensitivity; Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- test group-1- 10% propolis (Experimental): 10% propolis desensitizer, a pea-sized quantity was smeared over the test tooth. Subsequently, Iontophoresis was applied immediately. The desensitizing agent was administered at two intervals, immediately after oral prophylaxis and at the 14th-day visit.
  Interventions: Combination Product: desensitizing agents -10% Propolis
- test group -2- 2% sodium fluoride (Active Comparator): 2% sodium fluoride desensitizer, a pea-sized quantity was smeared over the test tooth. Subsequently, Iontophoresis was applied immediately. The desensitizing agent was administered at two intervals, immediately after oral prophylaxis and at the 14th-day visit.
  Interventions: Combination Product: desensitizing agents -10% Propolis
- test group-3- 1.23% acidulated phosphate fluoride (Active Comparator): 1.23% acidulated phosphate fluoride desensitizer, a pea-sized quantity was smeared over the test tooth. Subsequently, Iontophoresis was applied immediately. The desensitizing agent was administered at two intervals, immediately after oral prophylaxis and at the 14th-day visit.
  Interventions: Combination Product: desensitizing agents -10% Propolis

INTERVENTIONS:
Combination Product: desensitizing agents -10% Propolis — 10% propolis was prepared after mixing with 70% ethanol and distilled water based on the method described previously. Propolis and ethanol mixture was allowed to stay in dark place for two weeks. The mixture was stirred everyday intermittently for two weeks. Later the mixture was strained twice using filter paper to remove impurities.
  Propolis in general are fairly stable without losing its antibacterial properties for over 12 months when stored without direct sunlight and at cool temperatures. Alcohol based extracts will have extended shelf life and hence ethanol-extracted propolis prepared was stored in dark amber colored bottle without any preservatives.

SUMMARY:
Fluoridated desensitizers the frequently used for the treatment of dentin hypersensitivity (DH) with Iontophoresis. This study aimed to evaluate and compare the immediate and long-term effects of 10% Propolis with 2% sodium fluoride and 1.23% acidulated phosphate fluoride when applied along with Iontophoresis for the treatment of cervical dentin hypersensitivity (DH). Single-center, parallel, and double-blinded randomized clinical trials were conducted on systemically healthy patients, complaining about DH, with at least two sites. 10% propolis, 2% Sodium Fluoride and 1.23% Acidulated Phosphate Fluoride were used as desensitizers along with the Iontophoresis. After applying specific stimuli any decrease in DH was measured at baseline before and after application, on the 14th day after use, and at 28th-day post-intervention time intervals.

DETAILED DESCRIPTION:
Preparation of the materials 10 milligrams of Sodium Fluoride powder was mixed with 500 ml of distilled water to attain 500 ml of 2% concentrated Sodium Fluoride solution. Commercially available Acidulated Phosphate Fluoride was used at 1.23% concentration. Preparation of propolis: Commercially available raw Indian propolis in wax form was obtained from Hi-Tech Natural Product India Limited, New Delhi, India. 10% propolis was prepared after mixing with of 70% ethanol and distilled water based on the method described previously. Propolis and ethanol mixture was allowed to stay in a dark place for two weeks. The mixture was stirred everyday intermittently for two weeks. Later the mixture was strained twice using filter paper (Whatman International Ltd. England) to remove impurities. Propolis in general is fairly stable without losing its antibacterial properties for over 12 months when stored without direct sunlight and at cool temperatures. Alcohol-based extracts will have extended shelf life and hence ethanol-extracted propolis prepared was stored in the dark amber-colored bottle without any preservatives.

Study Design The trial was designed after multiple discussions among the authors and strictly followed the guidelines of CONSORT (Consolidated standards of reporting trials). It was a single centered, parallel, and double-blinded randomized clinical trial, approved by an institutional ethical review board and thesis protocol was registered in concerned medical university. Centralized computer-generated randomization was done without any restrictions. Randomization codes were kept sealed and managed by the central pharmacy to follow the allocation concealment. The DH measurements were performed by two blinded examiners (NMB and NRR), and averages were noted at each time interval. Each time, while checking, a new sheet of paper was given to the examiners to record the measurements, and to hide the old measures, to prevent bias. Interventions were carried out by another blinded author (TS). Cronbach's Alpha for inter-examiner reliability was found to be 0.92 and intra-examiner reliability 0.85 and 0.82 for examiner 1 and 2 respectively.

Study Participants Consecutive patients who visited the Department of Periodontology; from April 2019 to August 2020, with the DH as a chief complaint, with an age range of 25-60 years were invited to join in the study. Participating in the study was purely voluntary. Written informed consent was taken from each patient. The willing patients were assessed for following the necessary eligibility criteria.

Patients included were: Systemically healthy (based on the medical and drug history.), needing oral prophylaxis with moderate calculus (subjects who have moderately poor oral hygiene and needs teeth cleaning), at least two non-adjacent hypersensitive teeth with Schiff scale score as >1 with air blast stimulus and availability of a minimum of 10 evaluable natural teeth excluding third molars. However, patients excluded were: Undergoing orthodontic therapy, undertreatment for DH/using desensitizing dentifrice, pregnant women, any history of periodontal treatment before three months, any history of asthma, allergic to honey bee products and pollen, teeth with dental caries, attrition, abrasion, erosion, and lack of vitality.

Patients were allocated to three test groups after randomization. Oral prophylaxis was done in all three groups; baseline DH levels were then evaluated.

Application of desensitizing agents Vaseline was generally applied all over the gingiva and mucosa with a cotton pellet to foil the soft tissues from any undesired effect. Desensitizers used in test groups were 10% Propolis, 2% Sodium Fluoride, and 1.23% Acidulated Phosphate Fluoride for the first, second, and third group, respectively. A respective desensitizer, the pea-sized quantity was smeared over the test tooth. Subsequently, Iontophoresis was applied immediately in all three groups. The desensitizing agent was administered at two intervals, immediately after oral prophylaxis and at the 14th-day visit.

Application of Iontophoresis Iontophoresis equipment (Medical S.R.L., Italy) was used in this study. The procedure includes application of electric current on the test tooth for penetration of ions through dentinal tubules. Based on the patient arch size, the corresponding tray size is selected. A sponge used over the tray for placing the desensitizer. A particular desensitizer is applied in the sponge based on the respective subject's study group. The tray along with a sponge is then positioned in the patient mouth. The patient was instructed to hold the positive electrode of the iontophoresis unit with his/her palm. The negative electrode was connected to the metal plate in the tray. The unit is now switched on, and a current of 2 milliamperes is applied for one minute, based on manufacturer specifications. After one minute, the unit is switched off, and the same procedure is employed on the opposing arch. The patient is advised not to drink/eat or rinse his mouth for another half an hour.

Assessing clinical parameters Tactile, air blast and cold water stimuli were applied in the given order. Reduction of the DH (primary outcome) was traced at the baseline, immediately after ultrasonic scaling, and shortly after desensitizer application, postoperative 14 days before and after application of desensitizer, and postoperative 28 days without any application. A careful check for any adverse reactions with desensitizers was done at all intervals. The tactile test was done with the help of pressure sensitive probe. Immediate apical to the cementoenamel junction, the probe was moved from distal to mesial direction, graded as 1-10 on the visual analogue scale (VAS) based on the patient's discomfort. A four-graded Schiff's scale measured air stimulus. Zero was taken as no response, one as a response is noticed but the subject does not request for discontinuation of the stimulus, two as a response is noticed and the subject requests for discontinuation of the stimulus, three as pain is seen and the subject requests for discontinuation of the stimulus. A cold-water test was done with cold water application drop by drop with a disposable syringe, measured with VAS.

All the study subjects across study groups were provided with Colgate Regular Toothpaste and a soft-bristle toothbrush. The study subjects were demonstrated modified Stillman's toothbrushing technique on an oversized tooth model and instructed to brush once in the morning and once before sleep at night for 2-3 minutes from the first day till the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (based on the medical and drug history.), needing oral prophylaxis with moderate calculus (subjects who have moderately poor oral hygiene and needs teeth cleaning), at least two non-adjacent hypersensitive teeth with Schiff scale score as >1 with air blast stimulus and availability of a minimum of 10 evaluable natural teeth excluding third molars.

Exclusion Criteria:

* Undergoing orthodontic therapy, undertreatment for DH/using desensitizing dentifrice, pregnant women, any history of periodontal treatment before three months, any history of asthma, allergic to honey bee products and pollen, teeth with dental caries, attrition, abrasion, erosion, and lack of vitality.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
reduced dentin hypersensitivity | baseline (0 day) to 28th day
  significant reduction in dentin hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Raghavendra R Nagate, MDS, Principal Investigator — King Khalid University
Locations (1):
- College of Dentistry King Khalid University, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Purra AR, Mushtaq M, Acharya SR, Saraswati V. A comparative evaluation of propolis and 5.0% potassium nitrate as a dentine desensitizer: A clinical study. J Indian Soc Periodontol. 2014 Jul;18(4):466-71. doi: 10.4103/0972-124X.138695. PMID 25210261
- [Background] Torwane NA, Hongal S, Goel P, Chandrashekar BR, Jain M, Saxena E. A clinical efficacy of 30% ethenolic extract of Indian propolis and Recaldent in management of dentinal hypersensitivity: A comparative randomized clinical trial. Eur J Dent. 2013 Oct;7(4):461-468. doi: 10.4103/1305-7456.120675. PMID 24932122
- [Background] Madhavan S, Nayak M, Shenoy A, Shetty R, Prasad K. Dentinal hypersensitivity: A comparative clinical evaluation of CPP-ACP F, sodium fluoride, propolis, and placebo. J Conserv Dent. 2012 Oct;15(4):315-8. doi: 10.4103/0972-0707.101882. PMID 23112475